CLINICAL TRIAL: NCT06688604
Title: The Effect of Infant Attachment Barrier on Maternal Sadness and Adaptation: a Randomized Controlled Trial
Brief Title: The Effect of Mother-Infant Contact Barrier on Maternal Sadness and Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aysel Bulez, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-2022/14-21
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Mother Infant Contact
Keywords: Mother infant contact, contact barrier, maternal sadness, postpartum adaptation, midwifery,

STUDY DESIGN:
Intervention Model Description: Ensuring mother-infant skin-to-skin contact by the researcher within the first 5 minutes after cesarean and vaginal birth.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- vaginal birth (Experimental)
  Interventions: Behavioral: skin contact
- Childbirth with spinal and epidural anesthesia (Experimental)
  Interventions: Behavioral: skin contact
- Cesarean section under general anesthesia (No Intervention)

INTERVENTIONS:
Behavioral: skin contact — Ensuring mother-infant skin-to-skin contact by the researcher within the first 5 minutes after birth
  Arms: Childbirth with spinal and epidural anesthesia; vaginal birth

SUMMARY:
This study was conducted to investigate the effect of mother-infant contact deprivation on maternal sadness and maternal adaptation. The research is a randomized controlled experimental study. The intervention group consisted of mothers who had vaginal births or cesarean deliveries with epidural/spinal anesthesia (n: 198), while the control group included mothers who had cesarean deliveries under general anesthesia (n: 99). In the intervention group, mother-infant skin-to-skin contact was ensured within the first 10 minutes after birth. No intervention was made with the mothers in the control group. Both groups were assessed within the first 48 hours postpartum using the Mother-Infant Contact Barrier Scale, and on the 14th day postpartum, the Postpartum Self-Evaluation Scale and the Postpartum Maternal Sadness Evaluation Scale were administered to compare the results.

DETAILED DESCRIPTION:
This study was conducted to investigate the effect of mother-infant contact deprivation on maternal sadness and maternal adaptation. The research is a randomized controlled experimental study. The intervention group consisted of mothers who had vaginal births or cesarean deliveries with epidural/spinal anesthesia (n: 198), while the control group included mothers who had cesarean deliveries under general anesthesia (n: 99). In the intervention group, mother-infant skin-to-skin contact was ensured within the first 10 minutes after birth. No intervention was made with the mothers in the control group. Both groups were assessed within the first 48 hours postpartum using the Mother-Infant Contact Barrier Scale, and on the 14th day postpartum, the Postpartum Self-Evaluation Scale and the Postpartum Maternal Sadness Evaluation Scale were administered to compare the results.

ELIGIBILITY:
Inclusion Criteria:

Had given birth at Mardin Training and Research Hospital

* No physical and/or mental health issues
* No infectious diseases transmitted through contact
* Agreed to participate in the study
* Able to speak Turkish and/or does not have communication issues
* Single live birth with the baby
* Mothers who gave birth vaginally or via spinal anesthesia and had skin-to-skin contact with their baby within the first 5 minutes postpartum

Exclusion Criteria:

Foreign nationals, immigrants, or those with communication issues

* Individuals with any physical and/or mental health problems
* Those with infectious diseases transmitted through contact
* Individuals who did not agree to participate in the study
* Mothers whose baby was stillborn (ex) after birth
* Mothers whose babies were receiving treatment in the intensive care unit
* Those who do not wish to provide a phone number
* Women who gave birth vaginally or via spinal anesthesia and do not wish to establish contact with their baby
* Mothers who gave birth to twins or more babies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Maternal Sadness and Adaptation | 9 month
  The development, reliability and validity study of the scale was conducted by Küçük and Cesur (Küçük, E. (2022) Postpartum maternity blues assesment scale: Improvement, validity and reliability study) (Thesis No. 727989) [Master's thesis, Sivas Cumhuriyet University] National Thesis Center of the Council of Higher Education.) in 2022. The scale included questions prepared to determine the psychological changes that occur in the mother in the postpartum period and what kind of problems these changes may create in the mother. The scale was created as a 5-point Likert type to be answered by the participants. The scale contains 23 items. The items in the scale were applied as '1- Strongly disagree, 2-Disagree, 3-Undecided, 4-Agree, 5- Strongly Agree'. A high score on the scale indicates that the symptoms of maternal sadness in the postpartum period are high. A scale consisting of three sub-dimensions with 23 items (First Factor 'Maternal self-care dimension', second factor 'Infant care di
Postpartum Self-Assessment Scale | nine mounth
  It was decided to be developed by Lederman and Weingarten in 1981 to evaluate the adaptation process of women in the postpartum period to motherhood. It is a 4-point Likert-type scale with 82 items. There are 7 subscales that evaluate the Postpartum Self-Assessment Scale. Each subscale contains 10 to 13 items. 39 of the items in the scale are reverse-biased. The numbers of the reverse-biased items in the scale are as follows; 1, 2, 4, 6, 9, 10, 14, 15,16, 22, 29, 30, 32, 33, 36, 38, 40, 41, 42, 43, 44, 46, 47, 49, 51, 53, 54, 59, 61, 62, 67, 69, 71, 73, 77, 78, 79, 81, 82. The scale is measured with a 4-point assessment. Postpartum adjustment is evaluated based on the results of scores ranging from "1" to "4" (4: "Describes very much," 3: "Partially describes," 2: "Somewhat describes," 1: Does not describe at all"). Scoring for reverse items is done in the opposite way. The lowest possible score for the entire scale is 82, and the highest is 328. Low scores indicate that the adaptatio
Mother-Infant Contact Barrier Scale | nine mounth
  Development of the Scale and Examination of Its Psychometric Properties was conducted by Kömürcü Akik and Durak Batıgün (Akik, B. K., & Batıgün, A. D. (2020). Mother-Infant Contact Barrier Scale (ABTEÖ): Development and Psychometric Properties. Current Approaches in Psychiatry/Psikiyatride Guncel Yaklasimlar, 12.) in 2020. It was planned to be developed to measure possible contact barriers that may be experienced between the mother and the baby, such as difficulties in adaptation between the mother and the baby after birth and negative experiences related to birth, based on the mother's report. A total of 38-item question pool form was created by the authors. After the preliminary preparations, a 37-item form with Likert-type scores from 1 to 5 ("1 = Doesn't Apply to Me at All", "2 = Doesn't Apply to Me", "3 = Undecided", "4 = Applies to Me Somewhat", and "5 = Applies to Me Completely") was created. The 37-item version of the scale was applied to the participants. As a result of the v

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Training and research hospital, Mardin, artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eyquem A, de Saint Martin J. [Clinical significance of circulating autoantibodies]. Ann Immunol (Paris). 1977 Jan-Mar;128(1-2):285-6. French. PMID 322584
- [Background] Bystrova K, Ivanova V, Edhborg M, Matthiesen AS, Ransjo-Arvidson AB, Mukhamedrakhimov R, Uvnas-Moberg K, Widstrom AM. Early contact versus separation: effects on mother-infant interaction one year later. Birth. 2009 Jun;36(2):97-109. doi: 10.1111/j.1523-536X.2009.00307.x. PMID 19489802
- [Background] Rowe-Murray HJ, Fisher JR. Operative intervention in delivery is associated with compromised early mother-infant interaction. BJOG. 2001 Oct;108(10):1068-75. doi: 10.1111/j.1471-0528.2001.00242.x. PMID 11702839
- [Background] Karimi FZ, Sadeghi R, Maleki-Saghooni N, Khadivzadeh T. The effect of mother-infant skin to skin contact on success and duration of first breastfeeding: A systematic review and meta-analysis. Taiwan J Obstet Gynecol. 2019 Jan;58(1):1-9. doi: 10.1016/j.tjog.2018.11.002. PMID 30638460
- See also: WHO — https://www.who.int/publications/i/item/WHO-RHR-15.02